CLINICAL TRIAL: NCT05132270
Title: Efficacy and Safety of Combination of Hydroxyurea and Low-dose Thalidomide on Hemoglobin Synthesis in Thalassemia Patients
Brief Title: Clinical Experience of Thalidomide in Thalassemic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital Karachi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-0420
Record Dates: First submitted 2021-10-21; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Thalassemia, Beta
MeSH Terms: conditions — beta-Thalassemia | interventions — Hydroxyurea; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of hydroxyurea and thalidomide (Experimental): Hydroxyurea was continued at a dose of 10-20 mg/kg/day for 6 months and then thalidomide was added orally at a dose of 2-5mg/kg/day for 6 months.
  Interventions: Drug: hydroxyurea and thalidomide

INTERVENTIONS:
Drug: hydroxyurea and thalidomide — Evaluation of hydroxyurea and thalidomide combination use in beta-thalassemia patients

SUMMARY:
Objectives

Primary objective:

• To determine the efficacy and safety of the combination therapy of Hydroxyurea and thalidomide in beta-thalassemia patients.

Secondary objective:

• To determine the change in liver and spleen size of beta-thalassemia patients on the combination therapy

A single-arm non-randomized trial to evaluate the efficacy and safety of combination therapy of hydroxyurea and thalidomide in beta-thalassemia patients. It was a twelve months study. Participants were monitored for six months on Hydroxyurea alone and then the combination therapy of hydroxyurea and thalidomide for another six months. Findings of physical examination, vital signs, laboratory, and ultrasound findings were recorded at baseline, during and end of the study.

Sample Size and Population This study included 135 Beta-thalassemia patients.

DETAILED DESCRIPTION:
The purpose of the study was to evaluate the efficacy and safety of the combination therapy of hydroxyurea and thalidomide in beta-thalassemia patients. The participants were evaluated on the basis of eligibility criteria, consent was obtained and baseline investigations were performed on the screening visit. Participants were continued on Hydroxyurea (10-20mg/kg/day) for the first six months and then for the next six months thalidomide (2-5 mg/kg/day) was added to the intervention. Aspirin was also added (2-4mg/kg/day).

Efficacy:

Maintenance or rise in Hemoglobin (Hb) levels and changes in transfusion frequency before and after the use of combination therapy was used to evaluate the efficacy of the combination therapy. Good responders were the patients who were on transfusion and went off-transfusion after the combination therapy or individuals who were already off transfusion and after combination therapy demonstrated an increase in Hb of at least 1gm/dl. Responders were those who remained on transfusion on combination therapy but displayed a 50% reduction in blood requirements. Whereas, non-responders, were individuals who were off-transfusion before combination therapy and had improvement in Hb of <1gm/dl, or those who remained on transfusion during combination therapy and did not experience transfusion reduction of at least 50%.

Safety:

Safety of the drug was evaluated on the basis of the following parameters and intervention was discontinued or put on hold if:

* Creatinine >1.1mg/dl, Urea >43mg/dl),
* Liver function (SGPT >35mg/L)
* Absolute Neutrophil counts<2*109/L
* Platelets < 100*109/L

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical and genetic diagnosis of β-thalassemia major and intermedia
2. Patients who showed partial response or a decline in response to hydroxyurea
3. Patients who are not the candidates for the bone marrow transplant procedure.

Exclusion Criteria:

1. Married Patients
2. Patients with comorbidities such as liver, cerebrovascular, cardiovascular, or kidney diseases
3. Patients allergic to the drug ingredients
4. Patients with mental disorders
5. Patients who are enrolled in other clinical trials
6. Patients with a history of venous or arterial thrombosis

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in transfusion requirements | 6 months on combination therapy
  Change in transfusion needs (measured as blood volume in ml) per month from baseline
Change in Hemoglobin levels | 6 months on combination therapy
  Change in hemoglobin level of >1g/dl from baseline
Change in the liver function test | 6 months on combination therapy
  Change in SGPT in U/l from baseline
Change in liver function test | 6 months on combination therapy
  Change in total, direct, and indirect bilirubin in mg/dl from baseline
Change in Kidney Function test | 6 months on combination therapy
  Change in urea and creatinine levels in mg/dl from baseline

SECONDARY OUTCOMES:
Change in Spleen size | 6 months on combination therapy
  Change in size of spleen (in centimeters) from baseline
Change in liver size | 6 months on combination therapy
  Change in size of liver (in centimeters) from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ansari SH, Ansari I, Wasim M, Sattar A, Khawaja S, Zohaib M, Hussain Z, Adil SO, Ansari AH, Ansari UH, Farooq F, Masqati NU. Evaluation of the combination therapy of hydroxyurea and thalidomide in beta-thalassemia. Blood Adv. 2022 Dec 27;6(24):6162-6168. doi: 10.1182/bloodadvances.2022007031. PMID 35477175